CLINICAL TRIAL: NCT07007689
Title: A Multi-omics Study of BRAF V600E Mutant Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2025ZSLYEC-156
Record Dates: First submitted 2025-04-27; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: BRAF V600E-mutant Metastatic Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The fresh tumor tissues/biopsies and peripheral blood samples of each patient will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BRAF V600E mutant colorectal cancer cohort: Single-cell RNA sequencing, TCR sequencing, proteomics and metabolomics of 200 prospectively collected tissue samples. TCR sequencing of 200 prospectively collected blood samples.

SUMMARY:
This trial aims to elucidate the immune landscape and genetic basis of BRAF-mutant colorectal cancer (CRC) in Chinese patients by analyzing tumor tissue and peripheral blood. Single-cell RNA sequencing, T cell receptor (TCR) sequencing, proteomics and metabolomics, will be performed on tumor tissues, alongside TCR sequencing of peripheral blood, to establish a comprehensive immune and genetic profile of BRAF-mutant CRC. The study seeks to identify novel immune biomarkers, therapeutic targets, and signaling pathways, and to enable molecular subtyping for precision treatment and personalized management of BRAF-mutant CRC patients.

DETAILED DESCRIPTION:
As an oncogenic gene, BRAF V600E subverts the need for continuous upstream activation and overcomes negative feedback signals that terminate pathway activation. In colorectal cancer, BRAF V600E mutations are associated with older age, right colon primary tumors and female gender, as well as reduced chemotherapy sensitivity and poor prognosis. In addition to a poor prognosis, BRAF V600E-mutant colorectal cancer is associated with a higher incidence of peritoneal metastasis, resulting in tumor-related symptoms such as pain, ascites, gastrointestinal and urinary obstruction, which severely compromise patients' quality of life. Although there is a trend that BRAF V600E mutant patients who receive high-intensity chemotherapy have longer progression-free survival (PFS), the prognosis of the BRAF V600E mutant population remains dismal and approximately 40% of patients do not respond to first-line high-intensity chemotherapy. In addition, the response rate of combined targeted therapy is limited to around 25% and the duration of anti-epidermal growth factor receptor (EGFR) and anti-BRAF is around 4 months due to the presence of bypass activation. What's more, patients with BRAF V600E mutation and mismatch repair-proficient (pMMR) also had a poor response to anti-programmed death-1 (PD-1) therapy. The tumor heterogeneity and tumour immune microenvironment of BRAF V600E mutant colorectal cancer need to be investigated. The study seeks to identify novel immune biomarkers, therapeutic targets, and signaling pathways, and to enable molecular subtyping for precision treatment and personalized management of BRAF-mutant CRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to study procedures;
2. Men and women aged ≧18 years;
3. Diagnosis of histologically or cytologically confirmed colorectal cancer;
4. First-generation sequencing or next-generation sequencing at any time prior to screening confirms the presence of BRAF V600E mutation in tumor tissue.

Exclusion Criteria:

1. Patients with serious heart disease, hypertension, cerebral hemorrhage or uncontrollable systemic diseases (such as: diabetes, hypertension, pulmonary fibrosis and acute pneumonia);
2. Women who are pregnant or nursing;
3. Unable to co-operate in sampling;
4. Received more than two prior regimens of systemic cancer therapy for colorectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must meet all inclusion and exclusion criteria. In addition, the patient should be thoroughly informed about the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent. The written informed consent should be obtained from the patient prior toenrollment. The following criteria apply to all patients enrolled onto the study unless otherwise specified.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
prediction accuracy of treatment response | through study completion, an average of 3 years
  We will use gene data and treatment response data of the patients to construct a prediction model, the accuracy of model to anticipating partial response of patients is the primary.

SECONDARY OUTCOMES:
prediction of accuracy of survival rate | through study completion, an average of 3 years
  We will use the gene data and follow-up data of the patients to construct a prediction model, the accuracy of model to anticipating the 3-year survival rate of patients is the secondary endpoint.

IPD SHARING:
Plan to Share IPD: No